CLINICAL TRIAL: NCT00097305
Title: Delving Intervention and Mindbody Integration
Brief Title: Body-Oriented Therapy for Sexual Abuse Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F31AT001053 (NIH)
Record Dates: First submitted 2004-11-19; First posted 2004-11-22 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2006-08

CONDITIONS: Child Abuse, Sexual; Post-Traumatic Stress Disorder; Dissociation
Keywords: Mental Health; Psychotherapy
MeSH Terms: conditions — Coitus; Stress Disorders, Post-Traumatic; Dissociative Disorders; Psychological Well-Being

INTERVENTIONS:
Behavioral: Body-Oriented Therapy
Behavioral: Standardized Massage Therapy

SUMMARY:
The purpose of this study is to examine and compare the effects of two body therapy approaches in women who have experienced child sexual abuse.

DETAILED DESCRIPTION:
Women who have experienced child sexual abuse often display symptoms of dissociation and lack of bodily self-awareness which hinder the recovery process. Mind-body researchers have examined alternative therapeutic approaches to eliminating these factors. This study will compare a standardized therapeutic message to body-oriented therapy which involves a combination of hands-on bodywork and verbal therapy focused on somatic and emotional awareness.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported child sexual abuse
* In current psychotherapy for child sexual abuse recovery

Exclusion Criteria:

* Over 6 months of past experience with body-oriented therapy
* Diagnosis or medications for psychosis
* Drug or alcohol addiction
* Current abusive relationship
* Dissociative disorder
* In transition on psychotropic medication

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Price, PhD, Principal Investigator — Assistant Professor, University of Washington School of Nursing
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States

REFERENCES:
- [Background] Price, C. Characteristics of women seeking bodywork as an adjunct to psychotherapy during recovery from childhood sexual abuse. Journal of Bodywork and Movement Therapies, 8(1): 35-42, 2004.
- [Background] Price, C. Body-oriented therapy as an adjunct to psychotherapy in recovery from childhood abuse: A case study. Journal of Bodywork and Movement Therapies, 6(4): 228-236, 2002.
- [Background] Price C. Bodywork for childhood abuse treatment: a pilot-test comparison. 35th Annual Communicating Nursing Research Conference/16th Annual WIN Assembly, Health Disparities: Meeting the Challenge, April 18-20, 2002, Palm Springs, California. Communicating Nursing Research. 35(10):264, 2002.